CLINICAL TRIAL: NCT03071328
Title: INJECT: A Pilot Study of Intra-tumoral Injections in Metastatic Urological Cancers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00078508
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC); Metastatic Urothelial Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Bone metastatic site (Experimental)
  Interventions: Drug: Isovue-M 200
- Liver metastatic site (Experimental)
  Interventions: Drug: Isovue-M 200
- Lymph node metastatic site (Experimental)
  Interventions: Drug: Isovue-M 200
- Soft tissue metastatic site (Experimental)
  Interventions: Drug: Isovue-M 200

INTERVENTIONS:
Drug: Isovue-M 200 — Diluted iodinated contrast will be injected under CT fluoroscopy guidance into bone, lymph node, soft tissue, or liver metastases in subjects with metastatic castrate resistant prostate cancer, metastatic urothelial carcinoma or metastatic renal cell carcinoma and pre and post-injection CT images will be obtained to characterize the parameters needed for optimal distribution throughout metastases of a given size. To validate the expression of CD155 in prostate cancer, a biopsy of the metastatic site will be obtained at the time of contrast injection and will be stained for CD155 expression.
  Other Names: iodinated contrast

SUMMARY:
The purpose of this study is to plan for future clinical trials in patients with metastatic urological cancers. Diluted iodinated contrast will be injected intra-tumorally under CT fluoroscopy guidance into bone, lymph node, soft tissue and liver metastases in subjects with metastatic prostate cancer, urothelial carcinoma, or renal cell carcinoma. Pre- and post-injection CT images will be obtained to determine the injection parameters needed for optimal distribution throughout metastases of a given size. A biopsy of the metastatic site will also be obtained to validate expression of the receptor CD155.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate, renal cell carcinoma or urothelial carcinoma. Small cell or neuroendocrine tumors of the prostate are also permitted.
2. Radiographic evidence of at least one bone, lymph node, soft tissue, or liver metastasis, that is amenable to iodinated contrast injection, as judged by the study radiologist
3. Adequate laboratory values:

   1. Platelets ≥ 100,000
   2. INR ≤ 1.3
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. History of intercurrent or past medical or psychiatric illness that would make participation in a research biopsy protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Cr >2.0
3. History of iodinated contrast allergy
4. For patients undergoing research only biopsy: Requirement for anticoagulation with heparin, low molecular weight heparin, clopidogrel, rivaroxaban, dabigatran, apixaban, warfarin, Aggrenox, fondaparux, ticagrelor, etc (aspirin and other NSAIDs are ok but should be held prior to biopsy in accordance with institutional standard of care)
5. Any other contraindication to CT with iodinated contrast, as CT with contrast will be used in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of iodinated contrast enhancement within the metastasis on post-injection CT | Day 1
Percentage of iodinated contrast enhancement within the metastasis on post-injection CT | Day 1

SECONDARY OUTCOMES:
Presence of tumor CD155 membrane expression in metastatic bone, liver, soft tissue or lymph node specimens. | Day 1
  IHC will be used to assess tumor CD155 membrane expression in metastatic bone, liver, soft tissue, or lymph node specimens.
Estimated percentage of tumor CD155 membrane expression in metastatic bone, liver, soft tissue, or lymph node specimens. | Day 1
  IHC will be used to assess tumor CD155 membrane expression in metastatic bone, liver, soft tissue, or lymph node specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Megan McNamara, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States